CLINICAL TRIAL: NCT03192462
Title: Tumor-Associated Antigen (TAA) Specific Cytotoxic T Lymphocytes Administered in Patients With Pancreatic Cancer
Brief Title: TAA Specific Cytotoxic T Lymphocytes in Patients With Pancreatic Cancer
Acronym: TACTOPS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other); Pancreatic Cancer Action Network (Other); The V Foundation for Cancer Research (Other); Harris County Hospital District (Other Government)
Responsible Party: Principal Investigator, Benjamin Leon Musher, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-40378 TACTOPS
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Immune-based therapies; CytotoxicT Lymphocytes
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is designed as a fixed-dose pilot study to evaluate the safety and feasibility and efficacy of up to 6 intravenous infusions of multiTAA-specific T cells in pancreas cancer patients with metastatic, locally advanced unresectable, or resectable disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (Closed to New Patient Enrollment) (Experimental): Patients with locally advanced or metastatic pancreatic adenocarcinoma who are responding following 3 cycles of first line chemotherapy will receive 6 infusions with a fixed dose of multiTAA specific T cells beginning on the 4th week of the 4th cycle of chemotherapy. MultiTAA T cell infusions will occur on day 21 (a chemotherapy "off" week) of each chemotherapy cycle starting on chemotherapy cycle 4.
  Interventions: Biological: multiTAA specific T cells
- Group B (Closed to New Patient Enrollment) (Experimental): Patients with locally advanced or metastatic pancreatic adenocarcinoma who have failed first line chemotherapy or are intolerant or ineligible to receive standard of care chemotherapy will be evaluated in the clinic and receive 6 infusions (administered at monthly intervals) with a fixed dose of multiTAA specific T cells.
  Interventions: Biological: multiTAA specific T cells
- Group C (Closed to New Patient Enrollment) (Experimental): Patients with resectable pancreatic adenocarcinoma following completion of neoadjuvant chemotherapy, radiotherapy or combination. These patients will receive 6 infusions with a fixed dose of multiTAA specific T cells. One infusion will occur 4 weeks prior to surgical resection (with an option to infuse up to one week earlier) and after the completion of all pre-operative chemotherapy and/or radiation. The subsequent 5 infusions will occur at monthly intervals beginning 8 weeks post-surgery. Following surgery all patients will additionally receive 3 months of standard of care (SOC) chemotherapy starting week 9 after surgery. Hence, SOC chemo will occur weeks 9-11, 13-15, and 17-19 post-surgery and multiTAA T cell infusions will occur at weeks 8, 12, 16, 20, and 24 post-surgery.
  Interventions: Biological: multiTAA specific T cells

INTERVENTIONS:
Biological: multiTAA specific T cells — Each patient will receive 6 infusions of multiTAA T cells at a fixed cell dose (1 x 10^7 cells/m2) at the times specified in the group description. The expected volume of infusion will be 1 to 10 cc.

SUMMARY:
Status - CLOSED TO PATIENT ENROLLMENT (CNPE)

Patients who have pancreatic cancer that has come back or has not gone away after treatment, including the standard treatment for this disease or patients who are not eligible for or have elected not to receive standard of care chemotherapy, and patients who will have surgery after treatment for pancreatic cancer are eligible for this study. This is a research study using special immune system cells called tumor-associated antigen (TAA)-specific cytotoxic T lymphocytes, a new experimental therapy.

The proteins that are targeted in this study are called tumor-associated antigens (TAAs). These are cell proteins that are specific to the cancer cell. They do not show, or they show up in low quantities, on normal human cells. In this study, five common TAAs will be targeted. They are called NY-ESO-1, MAGEA4, PRAME, Survivin and SSX2. On a different study, patients have been treated and so far this treatment has shown to be safe.

Investigators now want to try this treatment in patients with pancreatic cancer.

These TAA-specific cytotoxic T lymphocytes (TAA-CTLs) are an investigational product not approved by the Food and Drug Administration.

*Arm A and Arm B are closed to new patient enrollment.*

DETAILED DESCRIPTION:
Status - CLOSED TO PATIENT ENROLLMENT (CNPE)

The patient will give blood to make TAA-Specific cytotoxic T cells in a lab. These cells well be grown and frozen. If the TAA-Specific cytotoxic T cells can be made, the time from collection of the blood to manufacture of T cells for administration to the patient is about 1 to 2 months.

The cells will be infused by intravenous infusion (IV) into the patient over 1-10 minutes. The patient may be pre-treated with acetaminophen (Tylenol) and diphenhydramine (Benadryl). Acetaminophen (Tylenol) and diphenhydramine (Benadryl) are given to prevent a possible allergic reaction to the TAA-CTL administration.

Patients will be given up to six doses of TAA-CTLs at monthly intervals. The treatments will be given by the Center for Cell and Gene Therapy at Houston Methodist Hospital (HMH).

MEDICAL TESTS BEFORE TREATMENT:

* Physical exam.
* Blood tests to measure blood cells, kidney and liver function.
* Measurements of the patient's tumor by routine imaging studies and/or blood tests. The study will use the imaging study that was used before to follow the patient's tumor: CT, MRI, or PET.
* Blood test to check for pregnancy for female patients who can have children

MEDICAL TESTS DURING TREATMENT:

Standard medical tests will be conducted on the day of the second and subsequent infusions:

* Physical exams prior to each T cell infusion
* Blood tests to measure blood cells, kidney and liver function.

MEDICAL TESTS AFTER TREATMENT:

- Measurements the patient's tumor by routine imaging studies and/or blood tests done as per standard of care.

To learn more about the way the TAA-CTLs are working in patient's body, an extra 20-40 mL (4-8 teaspoons) of blood will be taken before the infusion, at Weeks 1 and 2 after each infusion and at weeks 4, 6 and 8 and months 3, 6, 9 and 12 after the last infusion. The blood may be drawn from a central line at the time of the patient's regular blood tests. Investigators will use this blood to see how long the TAA-CTLs last, and to look at the immune system response to the patient's cancer.

Study Duration: Patients will be active participants in this study for approximately one year after their last dose. Investigators will contact patients once a year for up to 4 additional years (total of 5 years follow-up) in order to evaluate disease response long-term.

*Arm A and Arm B are closed to new patient enrollment.*

ELIGIBILITY:
Status - CLOSED TO PATIENT ENROLLMENT (CNPE)

Inclusion Criteria:

PROCUREMENT:

1. Any patient with biopsy proven pancreatic adenocarcinoma.
2. Patients with life expectancy greater than or equal to 6 months.
3. Age greater than or equal to 18 years
4. Hgb greater than or equal to 7.0 g/dl (transfusions allowed)

TREATMENT:

1. Any patient with biopsy-proven pancreatic adenocarcinoma:

   Group A: Patients with locally advanced or metastatic adenocarcinoma who are responding (defined as stable disease or tumor volume reduction) following 3 cycles of first line chemotherapy

   Group B: Patients with locally advanced or metastatic adenocarcinoma who have failed first line chemotherapy or are intolerant, ineligible or unwilling to receive standard of care chemotherapy

   Group C: Patients with resectable pancreatic cancer who have completed planned neo-adjuvant chemotherapy, radiotherapy or combination
2. Patients must have measurable or evaluable disease per RECIST 1.1 criteria.
3. Patients with life expectancy greater than or equal to 12 weeks
4. Age greater than or equal to 18
5. Pulse oximetry of greater than 95 percent on room air in patients who previously received radiation therapy
6. Patients with an ECOG score of ≤ 2 or Karnofsky score of 50 or greater
7. Patients with bilirubin less than or equal to 2x upper limit of normal, AST less than or equal to 3x upper limit of normal, Hgb greater than or equal to 7.0 g/dl (transfusion allowed).
8. Patients with a creatinine less than or equal to 2x upper limit of normal for age
9. Patients should have been off other investigational therapy for one month prior to receiving treatment on this study.
10. For Groups B or C patients must be off conventional therapy for at least 1 week prior to receiving treatment on this study.
11. Informed Consent explained to, understood by and signed by patient. Patient given copy of informed consent.
12. Due to unknown effects of this therapy on a fetus, pregnant women are excluded from this research. The male partner should use a condom. Females of child-bearing potential must be willing to utilize one of the more effective birth control methods during the study unless female has had a hysterectomy or tubal ligation.

Exclusion Criteria:

PROCUREMENT:

1. Patients with severe intercurrent infection.
2. Patients with active HIV infection (can be pending at this time)

TREATMENT:

1. Patients with severe intercurrent infection.
2. Patients receiving systemic corticosteroids (Patients off steroids for at least 48 hours are eligible)
3. Pregnant
4. HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2025-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Leen, PhD, Principal Investigator — Baylor College of Medicine; Benjamin Musher, MD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Baylor Clinic, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Harris Health System - Smith Clinic, Houston, Texas

REFERENCES:
- [Derived] Musher BL, Vasileiou S, Smaglo BG, Robertson CS, Wu M, Wang T, Watanabe A, Kuvalekar M, Velazquez Y, Ketkar S, Doheyan TA, Papayanni PG, Shah A, Lapteva N, Grilley BJ, Van Buren G, Lulla PD, Heslop HE, Rooney CM, Brenner MK, Leen AM. Autologous multiantigen-targeted T cell therapy for pancreatic cancer: a phase 1/2 trial. Nat Med. 2026 Jan;32(1):258-269. doi: 10.1038/s41591-025-04043-5. Epub 2026 Jan 2. PMID 41482561

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Patients with locally advanced or metastatic pancreatic adenocarcinoma who are responding following 3 cycles of first line chemotherapy will receive 6 infusions with a fixed dose of multiTAA specific T cells beginning on the 4th week of the 4th cycle of chemotherapy. MultiTAA T cell infusions will occur on day 21 (a chemotherapy "off" week) of each chemotherapy cycle starting on chemotherapy cycle 4.
  multiTAA specific T cells: Each patient will receive 6 infusions of multiTAA T cells at a fixed cell dose (1 x 10^7 cells/m2) at the times specified in the group description. The expected volume of infusion will be 1 to 10 cc.
- Group B: Patients with locally advanced or metastatic pancreatic adenocarcinoma who have failed first line chemotherapy or are intolerant or ineligible to receive standard of care chemotherapy will be evaluated in the clinic and receive 6 infusions (administered at monthly intervals) with a fixed dose of multiTAA specific T cells.
  multiTAA specific T cells: Each patient will receive 6 infusions of multiTAA T cells at a fixed cell dose (1 x 10^7 cells/m2) at the times specified in the group description. The expected volume of infusion will be 1 to 10 cc.
- Group C: Patients with resectable pancreatic adenocarcinoma following completion of neoadjuvant chemotherapy, radiotherapy or combination. These patients will receive 6 infusions with a fixed dose of multiTAA specific T cells. One infusion will occur 4 weeks prior to surgical resection (with an option to infuse up to one week earlier) and after the completion of all pre-operative chemotherapy and/or radiation. The subsequent 5 infusions will occur at monthly intervals beginning 8 weeks post-surgery. Following surgery all patients will additionally receive 3 months of standard of care (SOC) chemotherapy starting week 9 after surgery. Hence, SOC chemo will occur weeks 9-11, 13-15, and 17-19 post-surgery and multiTAA T cell infusions will occur at weeks 8, 12, 16, 20, and 24 post-surgery.
  multiTAA specific T cells: Each patient will receive 6 infusions of multiTAA T cells at a fixed cell dose (1 x 10^7 cells/m2) at the times specified in the group description. The expected volume of infusion will be 1 to 10 cc.
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 13 | 12 | 12
Completed | 0 | 0 | 2
Not Completed | 13 | 12 | 10
Not completed — Death | 13 | 11 | 10
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 13 | 12 | 12 | 37
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [55 to 69] | 51.5 [44 to 67.5] | 65 [62.5 to 67] | 63 [50 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 8 | 20
  Male | 7 | 6 | 4 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 6
  Not Hispanic or Latino | 11 | 10 | 9 | 30
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 2 | 0 | 0 | 2
  White | 11 | 10 | 11 | 32
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment Related Serious Adverse Events
Description: To determine the safety of up to 6 intravenous infusions of multiTAA-specific T cells in pancreatic cancer patients with metastatic, locally advanced unresectable, or resectable disease.
Time Frame: 7 months
Population: Participants who received at least one infusion of multiTAA-specific T cells.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 13 | 12 | 12
Participants | 0 | 1 | 0

2. Primary Outcome: Number of Patients Who Received 6 Infusions of multiTAA-specific T Cells
Description: To determine the feasibility of completing a total of 6 intravenous infusions of multiTAA-specific T cells to pancreatic cancer patients with metastatic, locally advanced unresectable, or resectable disease
Time Frame: 6 months
Population: Participants who received at least one infusion of multiTAA-specific T cells.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 13 | 12 | 12
Participants | 9 | 2 | 4

3. Secondary Outcome: Progression Free Survival Using the Kaplan-Meier Method
Description: To evaluate the progression-free of patients after multiTAA-specific T cell infusions. Progression-free survival (PFS) was estimated using the Kaplan-Meier method and summarized with median survival times and 95% confidence intervals. PFS was defined as the time from the first infusion to the first occurrence of disease progression, relapse, or death from any cause. Patients without events were censored at the last follow-up date.
Time Frame: 5 years
Population: The analysis population includes all participants who received at least one infusion of multiTAA-specific T cells.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 13 | 12 | 12
months | 6.4 [2.4 to 9.5] | 2.2 [1.2 to 2.5] | 7.5 [2.6 to 39.7]

4. Secondary Outcome: Overall Survival Using the Kaplan-Meier Method
Description: To evaluate the overall survival of patients after multiTAA-specific T cell infusions. Overall survival (OS) was estimated using the Kaplan-Meier method and summarized with median survival times and 95% confidence intervals. OS was defined as the time from the first infusion to death from any cause. Patients without events were censored at the last follow-up date.
Time Frame: 5 years
Population: The analysis population includes all participants who received at least one infusion of multiTAA-specific T cells.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 13 | 12 | 12
months | 14.1 [3.6 to 15.4] | 4.4 [1.5 to 16.7] | 12.6 [4.5 to 45.9]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality data was collected for 5 years and Serious and Other (Not Including Serious) Adverse Events were collected 8 weeks after the last dosing of the drug, up to 9 months.
Description: Adverse event data collection is still ongoing and will be updated upon study completion to include any additional adverse event data.
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 13/13 | 11/12 | 10/12
Serious Adverse Events (participants affected / at risk) | 4/13 | 6/12 | 3/12
Other Adverse Events (participants affected / at risk) | 13/13 | 12/12 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=13) | Group B (N=12) | Group C (N=12)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify : Cholangitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify : Large bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify : Ventral hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders and administration site conditions) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders and administration site conditions) | 3 (3) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, specify : Biliary Tract Obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify : Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infections and infestations - Other, specify : E. coli bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify : Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify : Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=13) | Group B (N=12) | Group C (N=12)
Anemia (Blood and lymphatic system disorders) | 7 (20) | 6 (10) | 10 (33)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (3) | 2 (2) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 4 (4) | 6 (7)
Bloating (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify : Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify : Indigestion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify : Melena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (6) | 3 (3) | 6 (6)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3)
Chills (General disorders and administration site conditions) | 4 (4) | 0 (0) | 1 (1)
Edema face (General disorders and administration site conditions) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders and administration site conditions) | 1 (2) | 0 (0) | 1 (1)
Fatigue (General disorders and administration site conditions) | 6 (7) | 8 (13) | 5 (5)
Fever (General disorders and administration site conditions) | 1 (2) | 4 (4) | 2 (2)
Flu like symptoms (General disorders and administration site conditions) | 1 (1) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify : Body aches (General disorders and administration site conditions) | 0 (0) | 2 (2) | 0 (0)
Malaise (General disorders and administration site conditions) | 1 (1) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders and administration site conditions) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders and administration site conditions) | 0 (0) | 0 (0) | 2 (2)
Hepatobiliary disorders - Other, specify : Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 3 (4)
Alanine aminotransferase increased (Investigations) | 7 (19) | 3 (5) | 6 (8)
Alkaline phosphatase increased (Investigations) | 6 (17) | 6 (7) | 5 (6)
Aspartate aminotransferase increased (Investigations) | 6 (16) | 4 (8) | 6 (11)
Blood bilirubin increased (Investigations) | 3 (4) | 4 (6) | 3 (4)
Creatinine increased (Investigations) | 0 (0) | 1 (2) | 2 (3)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 0 (0) | 3 (4)
Platelet count decreased (Investigations) | 3 (6) | 3 (3) | 6 (9)
Weight loss (Investigations) | 0 (0) | 0 (0) | 3 (4)
White blood cell decreased (Investigations) | 6 (16) | 2 (3) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (15) | 6 (8) | 6 (17)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (5) | 1 (2) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (20) | 6 (9) | 9 (14)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (9) | 2 (2) | 8 (14)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 4 (6) | 3 (4) | 5 (11)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 3 (4) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify : Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify : Pulled muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify : Lightheadedness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (10) | 1 (1) | 3 (3)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify : Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify : Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify : Loss of eyelashes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify : Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 8 (18) | 6 (12) | 6 (10)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders - Other, specify : Pulmonary emboli (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT03192462/Prot_SAP_000.pdf